CLINICAL TRIAL: NCT01838408
Title: Randomized, Single Blinded Study of Proposed EZ2go Complete Bowel Cleansing System: Evaluation of Its Safety, Efficacy and Patient Tolerance Compared to LOSO Prep, an Over the Counter Laxative Kit for Colonoscopy Bowel Preparation
Brief Title: Evaluation of Proposed EZ2go Complete Bowel Cleansing System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Borland-Groover Clinic (Other)
Collaborators: Valley Medical Products, LLC is paying for the study and is the sponsor. The form would not go through with this listed. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Pro00008184
Record Dates: First submitted 2013-04-16; First posted 2013-04-24 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Screening Colonoscopy; Surveillance Colonoscopy; Colonoscopy
Keywords: screening colonoscopy; surveillance colonoscopy; colonoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EZ2go Complete (Experimental): EZ2go complete: Peg 3350, Magnesium Citrate and Simethicone
  Interventions: Other: Ez2go Complete
- LoSo Prep ™ (Active Comparator): LoSo Prep ™: Magnesium citrate and Bisacodyl
  Interventions: Other: LoSo Prep

INTERVENTIONS:
Other: Ez2go Complete — EZ2Go Complete
  Arms: EZ2go Complete
Other: LoSo Prep — LoSo Prep ™ Magnesium Citrate plus Bisacodyl Kit Study Arm
  Arms: LoSo Prep ™

SUMMARY:
This study aims to provide safety and efficacy data comparable to available over-the-counter bowel preparations prior to colonoscopy. While there are many bowel preparations available, most of them remain expensive and require prescription from a health provider. The investigators believe EZ2go Complete will provide a non-inferior colon cleansing in a more accessible way (over-the-counter).

To accomplish this goal, the investigators decided to evaluate the proposed EZ2go combination versus currently available over-the-counter bowel preparations. The investigators believe the EZ2go kit will not be inferior to current FDA approved over-the-counter bowel preparations.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for routine colorectal cancer screening or surveillance colonoscopy examinations.
* Male and Female participants 18 years of age and older.
* Female participants who are not pregnant or planning to become pregnant within the next 90 days, or are sterile or of non-childbearing potential.
* Negative urine test at the screening visit.
* Subject is able to read and understand the informed consent form and signs the informed consent form.

Exclusion Criteria:

* Contraindication to any of the bowel preparations being used in the study.
* Unable/unwilling to fill out patient questionnaires following procedure.
* Pregnant or lactating.
* Unwilling to perform indicated lab work.
* Lab results that would indicate stage 4-5 chronic kidney disease (GFR <30MI/min1.73 m2).
* Personal history of colorectal cancer.
* Personal history of colorectal or small bowel surgery.
* Participants have any condition that, in the investigators opinion, could interfere with the participation and completion of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Measurement of Efficacy | 24 hours
  The primary end point is efficacy of colonoscopy preparation measured by the Ottawa scale.

SECONDARY OUTCOMES:
Evaluate the safety | 2 weeks
  A basic metabolic panel will be drawn at baseline and after the bowel preparation is complete to evaluate for any electrolyte and renal disturbances.

CONTACTS AND LOCATIONS:
Locations (1):
- Borland-Groover Clinic, Jacksonville, Florida, United States

REFERENCES:
- See also: Related Info — http://www.borland-groover.com